CLINICAL TRIAL: NCT06548438
Title: The Impact of PDD During TURB for NMIBC: a Prospective Randomized Controlled Trial
Brief Title: The Impact of PDD During TURB for NMIBC
Acronym: TUR_BLUE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Photocure (Industry)
Responsible Party: Principal Investigator, Francesco Soria, Principal Investigator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDS01FS
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer
Keywords: TURB; re-TURB; photodynamic diagnosis-PDD; Hexvix
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. Randomization will be stratified based on the dedicated surgeon performing the procedure. Allocation will be at a 1:1 ratio between the two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photodynamic diagnosis using Hexvix (Experimental): Transurethral resection of the bladder (TURB) is performed using photodynamic diagnosis (PDD) which involves the of use the study drug (Hexvix) to allow for better visualisation and subsequent resection
  Interventions: Procedure: Transurethral resection of the bladder performed with PDD tecnique and Hexvix
- White light (No Intervention): Transurethral resection of the bladder (TURB) is performed using the standard white light procedure

INTERVENTIONS:
Procedure: Transurethral resection of the bladder performed with PDD tecnique and Hexvix — For the execution of PDD cystoscopy in blue light, it is necessary to use the study drug (Hexvix) which, after intravesical instillation, causes an accumulation of porphyrins in the lesions of the bladder wall at the intracellular level. The intracellular porphyrins are photoactive fluorescent compounds that emit red light when excited with blue light. Consequently, the preneoplastic and neoplastic lesions will emit a red luminescence against a blue background, allowing for better visualisation and subsequent resection.
  Arms: Photodynamic diagnosis using Hexvix

SUMMARY:
The goal of this clinical trial is to learn if photodynamic diagnosis (PDD) performed using violet light after intra-vesical instillation of hexaminolaevulinic acid (Hexvix 85mg/50ml) is more sensitive than the standard white light tecnique in detection of malignant bladder tumour.

Patients will be randomised to:

* Transurethral resection of the bladder (TURB) with a standard white light tecnique
* TURB with the PDD tecnique using the study drug Hexvix

DETAILED DESCRIPTION:
Non-muscle invasive pT1 high-grade (HG) bladder cancer (NIMBC) represents a challenge for the urologists due to its aggressive behavior, with a marked tendency to recur after transurethral resection of the bladder (TURB) and even progress to muscle-invasive disease. To limit the risk of upstaging and to provide more clinical information indispensable for the decision-making process, international guidelines strongly recommend a re-TURB to be performed within 2-6 weeks from the first resection in all pT1HG tumors. However, not all the published literature agrees on the value of re-TURB wich is also an invasive and morbid procedure, requires a general or locoregional anesthesia and, like all surgical procedure, it is not free of risks and complications. There is, therefore, an unmet need for improving the quality and completeness of TURB which may have an impact on the necessity of Re-TURB. It has been confirmed that fluorescence-guided biopsy and resection (photodynamic diagnosis-PDD) are more sensitive than conventional procedures for the detection of malignant tumours, particularly for CIS. PDD is performed using violet light after intra-vesical instillation of hexaminolaevulinic acid (Hexvix 85mg/50ml).To date, no randomized controlled trials (RCTs) have been conducted aiming to compare the completeness of TURB with PDD compared to TURB with standard white light (WL).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent per Good Clinical Practice and national regulations
* Age ≥ 18 years
* Patient planned for TURB for >1,5 cm suspected (with either abdomen ultrasound or flexible cystoscopy) primary bladder cancer. The cut-off of 1,5cm has been chosen to maximize the probability of enrolling high-risk patients and, consequently, to maximize the probability of performing the re-TURB.

Exclusion Criteria:

* Patients with history of recurrent NMIBC
* Patients with visible incomplete resection during primary TURB
* Patients with metastatic disease or with a preoperative CT scan highly suspected for MIBC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Residual disease and/or upstaging | 6 to 8 weeks from the intervention
  Compare the completeness of TURB with PDD vs TURB with WL in terms of proportion of patients with residual disease and/or upstaging at re-TURB

SECONDARY OUTCOMES:
Number of Participants diagnosed with malignant lesions | 6 to 8 weeks from the intervention
  Compare the detection of malignant lesions between PDD and WLC using high-definition (HD) equipment during both primary TURB and re-TURB
The European organization for reasearch and treatment of cancer quality of life questionnaire for patients with non-muscle invasive bladder cancern | from date of randomization until 20 weeks from randomization
  The scale range from 24 (better outcome) to 96 (worse outcome)
EQ-5D-5L | from date of randomization until 20 weeks from randomization
  The scale range from 5 (better outcome) to 25 (worse outcome)
EQ VAS | from date of randomization until 20 weeks from randomization
  A self-rating question of overall health status, measured on a 0 (worse outcome) to 100 (better outcome) visual analogue scale
Adverse events | from date of randomization until 20 weeks from randomization
  Assess treatment changes and adverse events associated with each technique

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Soria, Principal Investigator — AOU Città della Salute e della Scienza

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data requests should be submitted to the corresponding author for consideration. Access to deidentified participant data may be granted following review, after the publication of major results
Supporting Information: Study Protocol
Time Frame: Data will be available after 6 months from major results publication and for the following 5 years
Access Criteria: Data requests should be submitted to the corresponding author for consideration